CLINICAL TRIAL: NCT00439426
Title: An Open Label Study of First Line Chemotherapy With Xeloda in Combination With Cisplatin on Treatment Response in Patients With Metastatic Nasopharyngeal Cancer
Brief Title: A Study of Xeloda (Capecitabine) in Combination With XELOX (Oxaliplatin) in Patients With Metastatic Nasopharyngeal Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20508
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Oxaliplatin; Capecitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: capecitabine [Xeloda]

INTERVENTIONS:
Drug: Oxaliplatin — 130mg/m2 iv on day 1 of each 3 week cycle
Drug: capecitabine [Xeloda] — 1000mg/m2 po bid on days 1-14 of each 3 week cycle

SUMMARY:
This single arm study will assess the efficacy and safety of Xeloda + oxaliplatin when given as first line treatment for patients with metastatic nasopharyngeal cancer. Patients will receive Xeloda (1000mg/m2 bid orally from day 1 to day 14, followed by a rest period of 7 days) plus oxaliplatin (130mg/m2 iv infusion on day 1 of each 21 day cycle) for 6-8 cycles. The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* history of nasopharyngeal cancer and distant metastases;
* no previous chemotherapy in past 6 months;
* recovery from previous radiotherapy;
* ability to swallow and retain oral medication.

Exclusion Criteria:

* previous cytotoxic chemotherapy;
* radiotherapy within 4 weeks of treatment start;
* history of another malignancy within the last 5 years;
* clinically significant cardiac disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Event driven

SECONDARY OUTCOMES:
Time to disease progression or death, survival time, duration of response, complete response rate. | Event driven
AEs, laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Morocco (4):
  - Agadir
  - Casablanca
  - Marrakesh
  - Rabat